CLINICAL TRIAL: NCT06713486
Title: Efficacy of Self-titration of Ventilation in Overlap Syndrome (chronic Obstructive Pulmonar Disease + Sleep Apnea Syndrome ) with Dynamic Hyperinflation. EDIN-IDIN.
Acronym: EDIN-IDIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EDIN-IDIN
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIXED PRESSURE (Experimental): Home nocturnal therapy either at the fixed pressure obtained in the polysomnography for 28 days
  Interventions: Procedure: Dynamic pressure in Dreamstation AVAPS-AAM PhilipsRespironic® mode
- B (Active Comparator): Dynamic pressure in Dreamstation AVAPS-AAM PhilipsRespironic® mode for 28 days.
  Interventions: Procedure: Fixed pressure obtained in the polysomnography for 28 days

INTERVENTIONS:
Procedure: Fixed pressure obtained in the polysomnography for 28 days — home nocturnal therapy either at the fixed pressure obtained in the polysomnography for 28 days
  Arms: B
Procedure: Dynamic pressure in Dreamstation AVAPS-AAM PhilipsRespironic® mode — dynamic pressure in Dreamstation AVAPS-AAM PhilipsRespironic® mode (program B) for 28 days, using the apnea threshold obtained in the titration as the maximum EPAP pressure and adjusting the support pressure for inferred Vt to 8 ml/kg of ideal body weight. After the first 28 days, a polysomnography will be performed under therapy with the device, and the next morning, cycle ergometry will be conducted.
  Arms: FIXED PRESSURE

SUMMARY:
The combination of COPD and obstructive sleep apnea (OSA) can lead to undesirable interactions with the treatment approach. The investigators know that continuous positive airway pressure (CPAP) can increase dynamic hyperinflation in COPD patients, and in mechanical ventilation, the increase in PEEP can worsen dynamic hyperinflation. On the other hand, the team know that the severity of COPD obstruction and hyperinflation alter sleep efficiency, with periods of wakefulness during sleep, and during these periods, the patient would not have upper airway obstruction, which could affect the therapy they are receiving in CPAP mode for OSA. Moreover, it was observed that with greater hyperinflation, the rate of obstructive events decreases, dynamically affecting the ventilatory situation with upper airway resistance. Recent studies have determined the safety and efficacy of auto-adjusting systems in the treatment of overlap syndrome, which could be more adaptable to the changing pulmonary mechanics of these patients. Aerobic capacity is a good predictor to the health status in these patients and the investigators know it is reduced in patients with AOS, where CPAP treatment according to studies improves the peak VO2. Therefore, the objective is to compare a ventilation system with fixed pressures established through polysomnography in patients with overlap syndrome and dynamic hyperinflation to a dynamic ventilation system using the fixed pressure limits typically established, based on their impact on the aerobic capacity (peak VO2) of these patients after 1 month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stability of at least 4 weeks without hospital admission.
* Previously presented PCO2 > 52.
* Age between 50 and 80 years.
* Agree to participate in the study and sign the informed consent.
* Both sexes.

Exclusion Criteria:

* Refusal to participate in the study.
* Uncontrolled structural or coronary heart disease (no changes in medication in the last 15 days).
* LVEF < 45%.
* Central sleep apnea syndrome (≥ 50% central events).
* Uncontrolled pulmonary hypertension.
* Inability to perform the tests.
* Having had an exacerbation 4 weeks prior.
* Severe psychiatric illness.
* Cognitive impairment.
* Not speaking Spanish.
* Illiteracy.
* Active smoker (or < 6 months since quitting smoking).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 | 0,29 and 57 days.
  Peak VO2 as the primary variable obtained from cycle ergometry.

SECONDARY OUTCOMES:
VO2 max | 0,29 and 57 days.
  VO2 max as a secondary variable obtained from cycle ergometry
Anaerobic threshold | 0,29 and 57 days.
  Anaerobic threshold as a secondary variable obtained from cycle ergometry.
VE/VCO2 | 0,29 and 57 days.
  The slope of VE/VCO2 obtained from cycle ergometry and resting PEtCO2.
BODE INDEX. (body mass index,) | 0,29 and 57 days.
  Polysomnography
BODE INDEX. ( air-flow obstruction) | 0,29 and 57 days.
  Time in hypoventilation period both during wakefulness and sleep, and as a function of total sleep time.
BODE INDEX. (dyspnea, ) | 0,29 and 57 days.
  number of residual respiratory events, time in hypoventilation period both during wakefulness and sleep, and as a function of total sleep time.
BODE INDEX. (exercise capacity) | 0,29 and 57 days.

OTHER OUTCOMES:
Epworth scale | 0,29 and 57 days.
  Based on a scale of (0 to 24 points)
Analytical parameters | 0,29 and 57 days.
  CAT u/ml
Analytical parameters | 0,29 and 57 days.
  ProBNP pg/mL
Analytical parameters | 0,29 and 57 days.
  C-reactive protein mg/dL
Analytical parameters | 0,29 and 57 days.
  pH
Analytical parameters | 0,29 and 57 days.
  pO2 mmHg, pCO2 mmHg
Analytical parameters | 0,29 and 57 days.
  sHCO3 mmol/L
Analytical parameters | 0,29 and 57 days.
  SatO2 %

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Neumología. Hospital Universitario Virgen de la Arrixaca., Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No